CLINICAL TRIAL: NCT00000675
Title: A Phase I Study of the Safety and Pharmacokinetics of Recombinant Human CD4 Immunoglobulin (rCd4-IgG) Administered by Intravenous Bolus in Patients With AIDS and AIDS Related Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: ACTG 121; DO136g
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-01

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; IgG; Drug Evaluation; Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex; Carrier Proteins
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — CD4 Immunoadhesins

INTERVENTIONS:
Drug: CD4-IgG

SUMMARY:
To study the safety and pharmacokinetics (blood levels) of recombinant human CD4 immunoglobulin (rCd4-IgG) in patients with AIDS or AIDS related complex (ARC) who have failed or declined therapy with zidovudine (AZT). An additional goal of the study is to obtain a preliminary indication of the antiviral effects of Cd4-IgG in patients with AIDS or ARC.

Other approaches in addition to existing treatment of HIV infection need to be evaluated. One approach may be to block HIV infection by interrupting the assembly of the virus within the cell or the budding of virus from the membrane of the infected cell. In addition, blocking the attachment of HIV to its cellular receptor may offer another point of attack. HIV binds to the CD4 receptor on the target T4 lymphocyte and the envelope glycoprotein of the virus (gp120) is capable of high affinity binding to CD4. Any agent that prevents the attachment of gp120 to the CD4 receptor should be able to block virus transmission and spread. Recently, scientists have succeeded in producing highly purified recombinant soluble human CD4. Recombinant CD4 is capable of binding to HIV envelope protein (gp120) and inhibiting HIV infectivity in test tube studies. Potential therapeutic benefit in patients with HIV infection could be derived from either or both of these biologic effects. In order to extend the length of time that rCD4 stays in the body, the compound has been modified by combining it with a human immunoglobulin of the IgG1 class (IgG).

DETAILED DESCRIPTION:
Other approaches in addition to existing treatment of HIV infection need to be evaluated. One approach may be to block HIV infection by interrupting the assembly of the virus within the cell or the budding of virus from the membrane of the infected cell. In addition, blocking the attachment of HIV to its cellular receptor may offer another point of attack. HIV binds to the CD4 receptor on the target T4 lymphocyte and the envelope glycoprotein of the virus (gp120) is capable of high affinity binding to CD4. Any agent that prevents the attachment of gp120 to the CD4 receptor should be able to block virus transmission and spread. Recently, scientists have succeeded in producing highly purified recombinant soluble human CD4. Recombinant CD4 is capable of binding to HIV envelope protein (gp120) and inhibiting HIV infectivity in test tube studies. Potential therapeutic benefit in patients with HIV infection could be derived from either or both of these biologic effects. In order to extend the length of time that rCD4 stays in the body, the compound has been modified by combining it with a human immunoglobulin of the IgG1 class (IgG).

Each patient receives rCd4-IgG at a fixed dose level once weekly by intravenous bolus for 12 weeks. Four patients (two per center) are entered at each dose level starting with the lowest dose. Dose escalation proceeds until a maximum tolerated dose (MTD) is defined. AMENDED: Includes, as of 891201, an ancillary study entitled "A Study of Recombinant CD4-Immunoglobulin G (CD4-IgG) Levels in Cerebral Spinal Fluid after rCD4-IgG is Administered by Intravenous Bolus in Patients With AIDS and AIDS-Related Complex". This involves selected patients, at the discretion of the Investigator. AMENDED: 900110 To increase the dose and frequency of administration of rCD4-IgG, based on preliminary results of pharmacokinetic analyses from Phase I studies in humans. Each patient receives rCD4-IgG therapy at a fixed dose level 1x, 2x, or 3x weekly by intravenous bolus for 12 weeks. Follow-up is extended to 8 weeks. Total target accrual is 25 - 28 weeks. AMENDED: 900824 Extension of the Phase I study of the safety and efficacy of CD4-IgG in patients with HIV infection. Each patient receives one of two fixed doses by IV bolus injection twice per week for 12 weeks. 20 to 30 patients to be enrolled. Pharmacokinetics will be evaluated. Clinical safety and antiviral effects will be assayed.

ELIGIBILITY:
Inclusion Criteria

Patients must fulfill the following criteria:

* Diagnosis of AIDS or AIDS-related complex, according to CDC criteria, in previously documented HIV seropositive individuals.
* Failure to tolerate or respond to zidovudine (AZT) therapy for HIV infection or a decision to decline such therapy.
* Willingness to abstain from all other experimental therapy for HIV infection during study period.
* Life expectancy of at least 3 months.
* Patients must be able to sign a written informed consent form.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Serious active opportunistic infection or malignancies not specifically allowed.

Concurrent Medication:

Excluded:

* Oral or intravenous acyclovir for herpes.
* Zidovudine (AZT).
* Interferon.
* Corticosteroids.
* Nonsteroidal anti-inflammatory agents (NSAIDS).
* Intravenous acyclovir.
* Other known immunomodulatory agents.
* Other experimental therapy.

Patients with the following are excluded:

* Serious active opportunistic infection or malignancies not specifically allowed.

Prior Medication:

Excluded within 4 weeks of study entry:

* Zidovudine (AZT).
* Chemotherapy.
* Immunomodulatory agents.
* Other experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: L Corey, Study Chair; A Collier, Study Chair
Locations (2):
- United States (2):
  - Stanford Univ School of Medicine, Stanford, California
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Collier AC, Coombs RW, Katzenstein D, Holodniy M, Gibson J, Mordenti J, Izu AE, Duliege AM, Ammann AJ, Merigan T, et al. Safety, pharmacokinetics, and antiviral response of CD4-immunoglobulin G by intravenous bolus in AIDS and AIDS-related complex. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Oct 1;10(2):150-6. doi: 10.1097/00042560-199510020-00006. PMID 7552478
- [Background] Collier A, Katzenstein D, Coombs R, Holodniy M, Mordenti J, Arditti D, Ammann A, Merigan T, Corey L. Safety and pharmacokinetics of intravenous recombinant CD4 immunoadhesin (RCD4-IGG) (AIDS Clinical Trials Group Protocol 121). Int Conf AIDS. 1990 Jun 20-23;6(3):206 (abstract no SB480)